CLINICAL TRIAL: NCT00968318
Title: Excision of Strip of Deep Fascia to Reduce Seroma Formation and Extrusion of Tissue Expanders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Professor Adel Wilson, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Reduce seroma with expanders
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Seroma
Keywords: Tissue expander; seroma; extrusion; lymphatics; deep fascia; Rate of seroma formation after excision of strip of deep fascia
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rate of seroma formation (Other): Excision of strip of deep fascia was assessed regarding the rate of seroma formation with tissue expander insertion
  Interventions: Procedure: Excision of strip of deep fascia

INTERVENTIONS:
Procedure: Excision of strip of deep fascia — operative technique to excise deep fascia.

SUMMARY:
Tissue expansion has enjoyed a wide range of applications since the technique was popularized in the latter quarter of the last century. During the expansion process, subcutaneous fat liquefies, skin becomes thinner, muscles atrophy, blood inflow increases, and lymphatics get occluded. All these factors predispose to seroma formation and implant extrusion.

A similar problem occurred with lymphoedema patients, and one of the lines of treatment was creation of a connection to the deep lymphatics to facilitate absorption of accumulated fluid. The same principle is to be extrapolated to patients having tissue expanders inserted in the neck and limbs and its effect is to be noted on the incidence of seroma .

DETAILED DESCRIPTION:
The techniques of tissue expansion have been used for many years to expand normal skin adjacent to the site of a defect. Initially described by Neuman in 1953, it gained widespread popularity in the eighth decade of the last century after the work of Radovan, and has been progressively popular since.

The physiology of prolonged tissue expansion was not just a matter of stretching skin, but the actual formation of additional new skin which had all the attributes of the original tissue. Austad et al. postulated that tissue expansion caused a decrease in cell density in the basal layer of the skin and that cell density might regulate skin mitotic activity. A lower cell density resulted in a greater cell proliferation, resulting in growth of additional skin. Inflation of the tissue expander was found to cause a threefold elevation of epidermal mitotic activity within 24 hours, followed by a gradual return to normal baseline over 2 to 5 days. Conversely, deflation of the expander caused a transient decrease in epidermal mitotic activity. The increase in mitosis returned to normal 4 weeks after expansion.

The dermis and subcutaneous tissues were thinned as a result of tissue expansion leading to an overall decrease in tensile strength of the expanded skin (5-7) and this persisted 36 weeks after expansion. The subcutaneous layer of fat was intolerant to stretching causing significant thinning. With faster expansion, fat necrosis could be seen. Pressure necrosis on subcutaneous fat led to liquefaction and seroma formation. With progression of expansion compression of superficial lymphatics resulted in their occlusion and lymph accumulation. Furthermore, the muscle layer in pigs, which was similar to the platysmal layer in humans, tended to atrophy with maximal expansion. As expansion proceeded, there was an increase in the number and size of the blood vessels within flaps supplied by random-pattern vessels and, if present, axial vessels. These changes corresponded to the demonstrated increase in blood flow to expanded flaps. In the study by Saxby this lead to surviving lengths after expansion being 50 percent greater than the delayed controls, and nearly 150 percent greater than comparable flaps raised acutely.

These histologic and physiologic findings would explain the high incidence of seroma formation with tissue expanders especially those inserted in areas rich in subcutaneous fat, such as the neck and limbs. During the expansion process, subcutaneous fat liquefies, skin becomes thinner, muscles atrophy, blood inflow increases, and lymphatics get occluded. All these factors when coupled with the fact that mere presence of a foreign body incites fluid exudation would be a frank invitation for seroma formation and implant extrusion.

Reported rates of seroma varied in the literature between 5-18%. Its effect ranged from minor complications that that did not interrupt the expansion process or require any operative intervention (32%) up to major complications that required additional operative intervention (12%).

Opinions differed between authors regarding seroma prevention. Several authors omit use of drainage procedures to prevent infection. Others use closed suction drains but there was an increased risk of infection; and seromas tended to occur following their removal.

External filling ports might drain seromas through the entry port, but at the risk of increased infection rates (19). Over inflation of the expanders to obliterate any dead space came with the risk of overlying skin ischemia and necrosis.

As a projection to the hypothesis of Thompson on lymphoedema management, this study was performed to find the effect of opening new drainage channels between the superficial and deep lymphatics on the incidence of seroma formation.

ELIGIBILITY:
Inclusion Criteria:

* Tissue expanders in neck and limbs.

Exclusion Criteria:

* Tissue expanders in other parts of the body.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2006-05; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Reduction of seroma formation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adel Wilson, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Adler N, Dorafshar AH, Bauer BS, Hoadley S, Tournell M. Tissue expander infections in pediatric patients: management and outcomes. Plast Reconstr Surg. 2009 Aug;124(2):484-489. doi: 10.1097/PRS.0b013e3181adcf20. PMID 19644263